CLINICAL TRIAL: NCT00030615
Title: A Phase I Study Of The Toxicities, Biologic And Clinical Effects Of Daily 5 Aza 2'Deoxycytidine (DAC), NSC 127716 (IND 50733) For Four Weeks In Patients With Advanced Malignancies
Brief Title: Decitabine in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02727; OC-01-01; U01CA062505 (NIH); CDR0000069182 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2002-02-14; First posted 2003-01-27 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Male Breast Cancer; Recurrent Bladder Cancer; Recurrent Breast Cancer; Recurrent Melanoma; Stage III Melanoma; Stage IV Bladder Cancer; Stage IV Breast Cancer; Stage IV Melanoma; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Breast Neoplasms, Male; Urinary Bladder Neoplasms; Breast Neoplasms; Melanoma | interventions — Decitabine

ARMS (1):
- Treatment (decitabine) (Experimental): Patients receive decitabine IV over 30 minutes on days 1-5 weekly for 4 weeks. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of decitabine until the MTD is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.
  Interventions: Drug: decitabine; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: decitabine — Given IV
  Other Names: 5-aza-dCyd; 5AZA; DAC
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial is studying the side effects and best dose of decitabine in treating patients with advanced solid tumors that have not responded to previous treatment. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose of decitabine in patients with advanced solid tumors.

II. Determine the toxic effects of this drug in these patients. III. Determine the dose of this drug with biologic activity in these patients. IV. Determine the pharmacokinetics of this drug in these patients. V. Determine clinical response to this drug in these patients.

OUTLINE: This is a dose-escalation, multicenter study.

Patients receive decitabine IV over 30 minutes on days 1-5 weekly for 4 weeks. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of decitabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed at 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced metastatic solid tumor for which all standard therapy has failed, including, but not limited to the following:

  * Stage III or IV melanoma

    * Mucosal melanoma allowed
    * No resectable stage III melanoma
  * Bladder cancer
  * Breast cancer
* No active symptomatic CNS disease
* No radiographically evident cerebral edema
* Hormone receptor status:

  * Not specified
* Male or female
* Performance status - ECOG 0-1
* Hemoglobin at least 9.0 g/dL
* Platelet count at least 100,000/mm^3
* WBC at least 3,500/mm^3
* Absolute granulocyte count at least 1,500/mm^3
* No coagulation disorders
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT and SGPT less than 2.5 times ULN
* Hepatitis B surface antigen negative
* Hepatitis C antibody negative
* Creatinine no greater than 1.5 times ULN
* No major cardiovascular system illness
* No major respiratory system illness
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No major systemic infection
* At least 1 month since prior radiotherapy
* At least 1 month since any prior anticancer therapy or adjuvant therapy
* No other experimental treatment within 30 days prior to, during, and for 30 days after study therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2001-12; Primary Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose determined by dose-limiting toxicities graded according to CTC 2.0 toxicity criteria | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Weber, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States